CLINICAL TRIAL: NCT03357055
Title: Ketamine Reduces Tourniquet Pain In Patients Undergoing Lower Limb Surgery Under Spinal Anaesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Foo Li Lian (Other)
Responsible Party: Sponsor-Investigator, Dr Foo Li Lian, Anaesthesiologist, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NMRR-17-2459-34013.
Record Dates: First submitted 2017-11-15; First posted 2017-11-29 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Tourniquet Pain
Keywords: tourniquet, pain, ketamine
MeSH Terms: conditions — Pain | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine arm (Experimental): Ketamine group will receive an IV infusion of 0.25mg/kg of ketamine in a 10 ml syringe over 10 minutes starting 10 minutes before pneumatic tourniquet inflation. Throughout the procedure patients will receive 0.25mg/kg of ketamine infusion at 10ml/hour until the end of operation.
  Interventions: Drug: Ketamine
- Control arm (Placebo Comparator): Control group will receive an intravenous (IV) infusion of 10 ml of normal saline in a 10 ml syringe over 10 minutes starting 10 minutes before pneumatic tourniquet inflation. Throughout the procedure, patients will receive 10ml/hour normal saline infusion until the end of operation.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — IV infusion of 0.25mg/kg of ketamine over 10 minutes before pneumatic tourniquet inflation. Throughout procedure patient will receive 0.25mg/kg of ketamine infusion.
  Arms: Ketamine arm
Drug: Normal saline — Control group will receive an intravenous (IV) infusion of 10 ml of normal saline in a 10 ml syringe over 10 minutes starting 10 minutes before pneumatic tourniquet inflation. Throughout the procedure, patients will receive 10ml/hour normal saline infusion until the end of operation
  Arms: Control arm

SUMMARY:
A prospective, double blind, randomised controlled trial to evaluate the effect of ketamine in reducing tourniquet pain for patients undergoing lower limb surgery under spinal anaesthesia.

Secondary Objective To evaluate the effect of ketamine in attenuating TIH for patients undergoing lower limb surgery under spinal anaesthesia.

DETAILED DESCRIPTION:
Primary Objective To evaluate the effect of ketamine in reducing tourniquet pain for patients undergoing lower limb surgery under spinal anaesthesia.

Secondary Objective To evaluate the effect of ketamine in attenuating TIH for patients undergoing lower limb surgery under spinal anaesthesia.

This will be a prospective, double blind, randomised controlled trial by multiple operators, who are medical officers in the Department of Anaesthesia, University Malaya Medical Centre. 60 patients will be recruited into the study. All patients recruited will be subjected to standard dose of spinal anaesthesia and randomly assigned into 2 different groups.

Methodology Patients will be fasted for at least 6 hours prior to their surgery. Oral midazolam 7.5 mg will be given to healthy adult from age 18-60 and 3.75mg will be given to adult age range from 60-65years as premedication prior to sending patients to the operating theatre.

Patients will be randomly assigned by principal investigator into one of two groups by using computer generated randomized numbers:

1. Control group will receive an intravenous (IV) infusion of 10 ml of normal saline in a 10 ml syringe over 10 minutes start 10 minutes before pneumatic tourniquet inflation. Throughout procedure patient will receive 10ml/hour normal saline infusion until operation finish.
2. Ketamine group will receive an IV infusion of 0.25mg/kg of ketamine in a 10 ml syringe over 10 minutes start 10 minutes before pneumatic tourniquet inflation. Throughout procedure patient will receive 0.25mg/kg of ketamine infusion in a 10ml syringe running at 10ml/hour until operation finish.

The study drug will be prepared on the morning of surgery by the principal investigator and anaesthetists in charge of the case is blinded to the grouping and to the drug. Standard monitoring with continuous electrocardiography (ECG), non-invasive blood pressure (NIBP) monitoring and pulse oximetry will be used for all patients. IV access will be established and co-loading of IV Hartman's solution 10ml/kg will be given. A baseline blood pressure reading of systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and heart rate (HR) will be taken prior to spinal anaesthesia. Patients will receive a spinal anaesthesia under aseptic technique using a 25-27 gauge Pencan® spinal needle. They will be given a dose of heavy bupivacaine 0.5% 2.5mls with fentanyl 20mcg added into the solution.

A pneumatic tourniquet using will be applied to the lower limb and inflated at 250mmHg above the systolic blood pressure. No additional sedation will be given to the patient intra-operatively.

Pain score will be assessed by blinded investigator using the 100 mm visual analog scale for pain (VAS for pain). Pain score using the VAS of 0 mm to 100mm will be recorded before application of the tourniquet(baseline), immediately after application of the tourniquet and thereafter every 10 minutes. SBP, DBP, MAP and HR will also be recorded at 10 minute intervals after the start of tourniquet inflation. The VAS and the blood pressure will be recorded at 10 minutes interval until the first reading after tourniquet deflation.

During the study period, if the VAS for pain score exceeds 40mm or if the SBP is elevated more than 30%, a dose of IV fentanyl 0.5 mcg/kg will be administered as rescue analgesia at 5 minutes interval and it will be recorded. If more than 3 doses of fentanyl given, case will be dropped out and manage according to local protocol (convert to general anaesthesia). If the SBP is persistently elevated more than 30% after 3 doses of IV fentanyl, they will be given IV labetalol 2.5mg and converted to GA and they will be dropped out from the study.

Maximum duration of tourniquet inflation was 130 minutes, after which surgeon would be advised to momentarily deflate the tourniquet and the study would be ended.

Statistical Analysis Normally distributed continuous data will be analyzed using t-test while non-parametric data will be analyzed by Mann Whitney U test using IBM SPSS Statistic version 23. Categorical data will be analyzed with Chi-square test and its non-parametric equivalent, Fisher's Exact test where appropriate. A p value < 0.05 will be regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1. ASA I or II 2. Age between 18-65 years old undergoing lower limb surgeries under spinal anaesthesia with pneumatic tourniquet inflation time more than 60 minutes

Exclusion Criteria:

* 1. Allergic to ketamine 2. Patients who have any degree of heart block, cardiovascular diseases, uncontrolled hypertension, severe peripheral vascular disease, sickle cell disease, diabetes neuropathy, deep vein thrombosis and pulmonary embolism, liver and renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-13 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores among patients in ketamine group vs patients in saline group, for patients undergoing lower limb surgery under spinal anaesthesia. | Pain scores will be assessed at baseline and throughout tourniquet application, at 10 minute intervals until 10 minutes after tourniquet deflation.
  Pain Score of 10-30mm: Mild pain Pain Score of 40-60mm: Moderate pain Pain Score of 70-100mm: Severe pain

SECONDARY OUTCOMES:
Change in blood pressure in ketamine group vs saline group, for patients undergoing lower limb surgery under spinal anaesthesia. | SBP, DBP, MAP and HR will be assessed at baseline and throughout tourniquet application, at 10 minute intervals until 10 minutes after tourniquet deflation
  Systolic, Diastolic blood pressure, Mean arterial pressure, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Lian Foo, Principal Investigator — Anaesthesiologist, Department of Anaesthesia, University Malaya Medical Centre

IPD SHARING:
Plan to Share IPD: No